CLINICAL TRIAL: NCT03335696
Title: Predicting MRI Abnormalities With Longitudinal Data of the Whitehall II Substudy
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: MSD/IDREC/C1/2011/71
Record Dates: First submitted 2017-09-29; First posted 2017-11-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2017-11

CONDITIONS: Cognitive Impairment; Dementia; Affective Disorders
Keywords: Epidemiology; Magnetic resonance imaging; Diffusion tensor imaging; White matter; Functional MRI; Connectome; Resting state brain networks; Neuropsychology
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White cells, buccal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Follow-up study within the Whitehall II study, selecting 800 participants for further neuropsychological, clinical and imaging (MRI) examinations to examine brain structure and function in relation to age-related diseases and the modifiable and non-modifiable factors affecting resilience against and vulnerability to adverse brain changes.

DETAILED DESCRIPTION:
A total of 6035 civil servants participated in the WHII Phase 11 clinical examination in 2012-2013. A random sample of 800 of these participants was included in a sub-study comprising an MRI brain scan, a detailed clinical and cognitive assessment, and collection of blood and buccal mucosal samples for the characterisation of immune function and associated measures. Data collection for this sub-study started in 2012 and was completed by in 2016. The participants, for whom social and health records have been collected since 1985, were between 60-85 years of age at the time the MRI study started. The pre-specified clinical and cognitive assessment protocols, the state-of-the-art MRI sequences and latest pipelines for analyses of this sub-study have been published and are attached to this application.

ELIGIBILITY:
Inclusion Criteria:

* Member of Whitehall II cohort attending at UCL for phase 11

Exclusion Criteria:

* Not suitable for MRI, travelling to Oxford, seriously physically ill

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Randomly selected from phase 11 of the an occupational cohort recruited from 1985 for the Whitehall II study (Marmot M, Brunner E. Cohort Profile: the Whitehall II study. Int J Epidemiol 2005;34(2):251-6).
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Neuropsychological measure 1 | 2012-2016
  National Adult Reading Test (premorbid intellectual ability)
Neuropsychological measure 2 | 2012-2016
  Montreal Cognitive Assessment (MoCA)
Neuropsychological measure 3 | 2012-2016
  Rey Complex Figure copy and delayed recall (visual episodic memory)
Neuropsychological measure 4 | 2012-2016
  Hopkins Verbal Learning Test Revised (verbal episodic memory)
Neuropsychological measure 5 | 2012-2016
  CANTAB Simple and Choice Reaction Time (processing speed)
Neuropsychological measure 6 | 2012-2016
  WAIS-R Digit Symbol Test (processing speed)
Neuropsychological measure 7 | 2012-2016
  Trail Making Test A and B (processing speed/executive functioning)
Neuropsychological measure 8 | 2012-2016
  WAIS-R Digit Span forward and backwards (executive functioning)
Neuropsychological measure 9 | 2012-2016
  Graded Naming Test (semantic memory)
MRI Measures 1 | 2012-2016
  Siemens 3T - T1-weighted scan (MPRAGE) using FSL FIRST, FAST, and Freesurfer Volume extractions
MRI Measures 2 | 2012-2016
  Siemens 3T - T1-weighted scan (MPRAGE) using FSL GLM Voxel based analysis for grey matter density analysis
MRI Measures 3 | 2012-2016
  Siemens 3T - T2-weighted scan, clinical and FSL (BIANCA)-based rating of white matter changes
MRI Measures 4 | 2012-2016
  Siemens 3T Diffusion Tensor Images analyzed with Tract Based Spatial Statistics (TBSS)
MRI Measures 5 | 2012-2016
  Siemens 3T rs-fMRI analyzed with Multivariate Exploratory Linear Optimized Decomposition into Independent Components: MELODIC)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus P Ebmeier, MD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study follows MRC data sharing policies. Data will be accessible from the authors after 2019.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After 2019
Access Criteria: approval by data sharing committee
URL: https://www.mrc.ac.uk/research/policies-and-guidance-for-researchers/data-sharing/

REFERENCES:
- [Result] Filippini N, Zsoldos E, Haapakoski R, Sexton CE, Mahmood A, Allan CL, Topiwala A, Valkanova V, Brunner EJ, Shipley MJ, Auerbach E, Moeller S, Ugurbil K, Xu J, Yacoub E, Andersson J, Bijsterbosch J, Clare S, Griffanti L, Hess AT, Jenkinson M, Miller KL, Salimi-Khorshidi G, Sotiropoulos SN, Voets NL, Smith SM, Geddes JR, Singh-Manoux A, Mackay CE, Kivimaki M, Ebmeier KP. Study protocol: The Whitehall II imaging sub-study. BMC Psychiatry. 2014 May 30;14:159. doi: 10.1186/1471-244X-14-159. PMID 24885374
- [Result] Allan CL, Zsoldos E, Filippini N, Sexton CE, Topiwala A, Valkanova V, Singh-Manoux A, Tabak AG, Shipley MJ, Mackay C, Ebmeier KP, Kivimaki M. Lifetime hypertension as a predictor of brain structure in older adults: cohort study with a 28-year follow-up. Br J Psychiatry. 2015 Apr;206(4):308-15. doi: 10.1192/bjp.bp.114.153536. Epub 2014 Dec 11. PMID 25497301
- [Result] Topiwala A, Allan CL, Valkanova V, Zsoldos E, Filippini N, Sexton CE, Mahmood A, Singh-Manoux A, Mackay CE, Kivimaki M, Ebmeier KP. Resilience and MRI correlates of cognitive impairment in community-dwelling elders. Br J Psychiatry. 2015 Nov;207(5):435-9. doi: 10.1192/bjp.bp.114.152363. Epub 2015 Sep 3. PMID 26338988
- [Result] Allan CL, Sexton CE, Filippini N, Topiwala A, Mahmood A, Zsoldos E, Singh-Manoux A, Shipley MJ, Kivimaki M, Mackay CE, Ebmeier KP. Sub-threshold depressive symptoms and brain structure: A magnetic resonance imaging study within the Whitehall II cohort. J Affect Disord. 2016 Nov 1;204:219-25. doi: 10.1016/j.jad.2016.06.049. Epub 2016 Jun 21. PMID 27372409
- [Result] Griffanti L, Jenkinson M, Suri S, Zsoldos E, Mahmood A, Filippini N, Sexton CE, Topiwala A, Allan C, Kivimaki M, Singh-Manoux A, Ebmeier KP, Mackay CE, Zamboni G. Classification and characterization of periventricular and deep white matter hyperintensities on MRI: A study in older adults. Neuroimage. 2018 Apr 15;170:174-181. doi: 10.1016/j.neuroimage.2017.03.024. Epub 2017 Mar 15. PMID 28315460
- [Result] Suri S, Emir U, Stagg CJ, Near J, Mekle R, Schubert F, Zsoldos E, Mahmood A, Singh-Manoux A, Kivimaki M, Ebmeier KP, Mackay CE, Filippini N. Effect of age and the APOE gene on metabolite concentrations in the posterior cingulate cortex. Neuroimage. 2017 May 15;152:509-516. doi: 10.1016/j.neuroimage.2017.03.031. Epub 2017 Mar 18. PMID 28323160
- [Result] Topiwala A, Allan CL, Valkanova V, Zsoldos E, Filippini N, Sexton C, Mahmood A, Fooks P, Singh-Manoux A, Mackay CE, Kivimaki M, Ebmeier KP. Moderate alcohol consumption as risk factor for adverse brain outcomes and cognitive decline: longitudinal cohort study. BMJ. 2017 Jun 6;357:j2353. doi: 10.1136/bmj.j2353. PMID 28588063
- [Result] Sexton CE, Zsoldos E, Filippini N, Griffanti L, Winkler A, Mahmood A, Allan CL, Topiwala A, Kyle SD, Spiegelhalder K, Singh-Manoux A, Kivimaki M, Mackay CE, Johansen-Berg H, Ebmeier KP. Associations between self-reported sleep quality and white matter in community-dwelling older adults: A prospective cohort study. Hum Brain Mapp. 2017 Nov;38(11):5465-5473. doi: 10.1002/hbm.23739. Epub 2017 Jul 26. PMID 28745016
- [Result] Suri S, Topiwala A, Filippini N, Zsoldos E, Mahmood A, Sexton CE, Singh-Manoux A, Kivimaki M, Mackay CE, Smith S, Ebmeier KP. Distinct resting-state functional connections associated with episodic and visuospatial memory in older adults. Neuroimage. 2017 Oct 1;159:122-130. doi: 10.1016/j.neuroimage.2017.07.049. Epub 2017 Jul 26. PMID 28756237
- [Result] Heise V, Zsoldos E, Suri S, Sexton C, Topiwala A, Filippini N, Mahmood A, Allan CL, Singh-Manoux A, Kivimaki M, Mackay CE, Ebmeier KP. Uncoupling protein 2 haplotype does not affect human brain structure and function in a sample of community-dwelling older adults. PLoS One. 2017 Aug 3;12(8):e0181392. doi: 10.1371/journal.pone.0181392. eCollection 2017. PMID 28771482
- [Derived] Patel R, Mackay CE, Jansen MG, Devenyi GA, O'Donoghue MC, Kivimaki M, Singh-Manoux A, Zsoldos E, Ebmeier KP, Chakravarty MM, Suri S. Inter- and intra-individual variation in brain structural-cognition relationships in aging. Neuroimage. 2022 Aug 15;257:119254. doi: 10.1016/j.neuroimage.2022.119254. Epub 2022 Apr 28. PMID 35490915
- [Derived] Jansen MG, Griffanti L, Mackay CE, Anaturk M, Melazzini L, Lange AG, Filippini N, Zsoldos E, Wiegertjes K, Leeuw FE, Singh-Manoux A, Kivimaki M, Ebmeier KP, Suri S. Association of cerebral small vessel disease burden with brain structure and cognitive and vascular risk trajectories in mid-to-late life. J Cereb Blood Flow Metab. 2022 Apr;42(4):600-612. doi: 10.1177/0271678X211048411. Epub 2021 Oct 5. PMID 34610763
- [Derived] Suri S, Chiesa ST, Zsoldos E, Mackay CE, Filippini N, Griffanti L, Mahmood A, Singh-Manoux A, Shipley MJ, Brunner EJ, Kivimaki M, Deanfield JE, Ebmeier KP. Associations between arterial stiffening and brain structure, perfusion, and cognition in the Whitehall II Imaging Sub-study: A retrospective cohort study. PLoS Med. 2020 Dec 29;17(12):e1003467. doi: 10.1371/journal.pmed.1003467. eCollection 2020 Dec. PMID 33373359
- [Derived] Zsoldos E, Mahmood A, Filippini N, Suri S, Heise V, Griffanti L, Mackay CE, Singh-Manoux A, Kivimaki M, Ebmeier KP. Association of midlife stroke risk with structural brain integrity and memory performance at older ages: a longitudinal cohort study. Brain Commun. 2020 Mar 7;2(1):fcaa026. doi: 10.1093/braincomms/fcaa026. eCollection 2020. PMID 32954286
- See also: Whitehall Imaging Oxford — https://www.psych.ox.ac.uk/research/neurobiology-of-ageing/research-projects-1/whitehall-oxford